CLINICAL TRIAL: NCT00141609
Title: A Study Looking at the Effects of a Modest Reduction in Dietary Salt Intake on Blood Pressure Control in Haemodialysis Patients
Brief Title: Haemodialysis Salt Reduction Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St George's, University of London (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LREC 04.0013
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2007-05-14 (Estimated); Status verified 2007-05

CONDITIONS: Kidney Failure, Chronic; Hypertension
Keywords: End-stage renal failure; Haemodialysis; Sodium; Blood Pressure
MeSH Terms: conditions — Kidney Failure, Chronic; Hypertension

INTERVENTIONS:
Drug: Slow Sodium

SUMMARY:
High blood pressure (hypertension) affects up to 80% of all patients receiving haemodialysis for chronic kidney disease (CKD). High blood pressure is a major cause cardiovascular disease (i.e. strokes, heart attacks and heart failure) and, thereby, cardiovascular deaths in these patients.

A significant cause of raised blood pressure in haemodialysis patients is thought to be due to retention of salt in the body. In healthy people the kidneys excrete salt but the kidneys of patients with CKD cannot do this, so salt has to be removed by dialysis. However dialysis cannot remove as much salt as is necessary, and so it accumulates. This fact has been recognized for many years, and health professionals caring for haemodialysis patients often stress the importance of restriction of dietary salt intake.

However no research has looked in detail at the mechanisms by which salt raises blood pressure in haemodialysis patients. It is likely that salt directly affects thirst, causing patients to drink more and become overloaded with fluid. In addition, salt may have direct effects on the blood vessel wall, causing failure of adequate blood vessel relaxation. Both of these factors may raise blood pressure.

We will conduct a carefully controlled crossover study looking at the effects of a modest reduction in salt intake on BP. During the course of the study, which will last eight weeks, patients will receive both a 5 gram per day and a 10 gram per day salt intake. We will look at how thirst, fluid intake, a number of markers of blood vessel function and blood pressure differ on these two salt intakes.

DETAILED DESCRIPTION:
High blood pressure (BP) is a major independent risk factor for cardiovascular mortality in individuals on haemodialysis, and yet BP is extremely poorly controlled in this population.

Excessive dietary salt intake is likely to be a major cause of hypertension in these patients. Firstly, excessive salt intake will result in thirst, excessive fluid intake and weight gains between dialysis, and thereby chronic over-expansion of extracellular fluid volumes resulting in high blood pressure. Secondly, salt may have direct effects on the arterial tree contributing to endothelial dysfunction that has clearly been demonstrated in uraemic individuals, including haemodialysis patients. Abnormalities in endothelial nitric oxide (NO) production may play an important role in salt-sensitive hypertension, mediated by the potent inhibitor of NO synthase, asymmetrical dimethylarginine (ADMA). Plasma ADMA concentrations are several-fold higher in individuals on dialysis than in normal controls, and it would be of interest to see whether ADMA concentrations decrease with a reduction dietary salt intake.

In spite of the importance of dietary salt intake in haemodialysis patients, there are no controlled studies which delineate the mechanisms by which salt intake affects BP. We propose to conduct a prospective double-blind placebo controlled cross-over study of normal (10 to 12 grams salt per day) versus modestly reduced (6 grams per day) salt intake over an eight week period in haemodialysis patients. The primary outcome measure is the change in pre-dialysis systolic BP. Other outcome measures include mean systolic and diastolic BP as measured by ABPM, thirst scores, daily weight gains and thoracic fluid content, as measured by thoracic bioimpedance. Furthermore, in a sub-group of subjects will we study the changes in plasma ADMA concentrations with reductions in salt intake, and examine correlations with changes in BP and systemic vascular resistance.

ELIGIBILITY:
Inclusion Criteria:

* Haemodialysis/haemodiafiltration for ESRF for >3 months
* Clinically stable

Exclusion Criteria:

* Significant intercurrent illness
* Systolic BP >240 mmHg/diastolic BP >120 mmHg at enrollment
* Unstable blood pressure whilst on HD
* Sodium profiled haemodialysis/HDF

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2004-04; Study Completion 2006-10

PRIMARY OUTCOMES:
Change in pre-dialysis systolic blood pressure

SECONDARY OUTCOMES:
Change in post-dialysis ambulatory BP (24 hr)
Change in thirst score
Change in intra-dialytic weight gain
Change in systemic vascular resistance
Change in assymmetric dimethylarginine (ADMA)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy WR Doulton, MBBS BSc MRCP, Principal Investigator — SGUL
Locations (1):
- Blood Pressure Unit, Cardiac & Vascular Sciences, SGUL, London, United Kingdom

REFERENCES:
- [Derived] McMahon EJ, Campbell KL, Bauer JD, Mudge DW, Kelly JT. Altered dietary salt intake for people with chronic kidney disease. Cochrane Database Syst Rev. 2021 Jun 24;6(6):CD010070. doi: 10.1002/14651858.CD010070.pub3. PMID 34164803